CLINICAL TRIAL: NCT04281576
Title: A Phase 2, Single Arm, Multi-center, Open-Label Trial to Evaluate the Safety and Efficacy of Treatment with Tumor Treating Fields (TTFields) and Chemotherapy As First-Line Treatment for Subjects with Unresectable Gastroesophageal Junction (GEJ) Adenocarcinoma or Gastric (GC) Adenocarcinoma
Brief Title: Effect of Tumor Treating Fields (TTFields, 150 KHz) Concomitant with Chemotherapy As First Line Treatment of Unresectable Gastroesophageal Junction or Gastric Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF-31 / ZL-8301-001
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer
Keywords: TTFields; XELOX; Oxaliplatin; Capecitabine; Minimal toxicity; TTF; Tumor Treating Fields; Novocure; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- NovoTTF-100L(P) (Experimental): Patients receive TTFields using the NovoTTF-100L(P) System together with XELOX. For HER-2 positive patients, Trastuzumab is given together with XELOX.
  Interventions: Device: NovoTTF-100L(P); Drug: Oxaliplatin; Drug: Capecitabine; Drug: Trastuzumab

INTERVENTIONS:
Device: NovoTTF-100L(P) — Patients receive continuous TTFields treatment using the NovoTTF-100L(P) device. TTFields treatment will consist of wearing four electrically insulated electrode arrays on the abdomen. The treatment enables the patient to maintain regular daily routine.
  Other Names: TTFields
Drug: Oxaliplatin — Oxaliplatin 130 mg/m^2 intravenous infusion will be administered once every 3 weeks
  Other Names: Eloxatin
Drug: Capecitabine — Capecitabine 1000mg/m^2 taken by mouth, twice daily on day 1-14, 3 weeks per cycle
  Other Names: Xeloda
Drug: Trastuzumab — Trastuzumab (HER-2 positive patients only) intravenous infusion will be administered once every 3 weeks on Day 1 of each cycle. First dose is 8mg/kg, followed by 6 mg/kg.
  Other Names: Herceptin

SUMMARY:
The study is a prospective, single arm, phase II trial aimed to evaluate the efficacy and safety of Tumor Treating Fields (TTFields) concomitant with XELOX for the treatment of unresectable, locally advanced or metastatic Gastroesophageal Junction (GEJ) or Gastric (GC) Adenocarcinoma who were previously untreated with systemic therapy. The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE-CLINICAL AND CLINICAL EXPERIENCE:

The effect of the electric fields (TTFields, TTF) has demonstrated significant activity in in vitro gastric cancer pre-clinical models both as a single modality treatment and in combination with chemotherapies. In addition, TTFields have shown to inhibit metastatic spread of malignant melanoma in in vivo experiment.

Prospective, multi-center clinical studies of TTFields have shown the safety of the treatment when administered to the abdomen for pancreatic cancer and ovarian cancer.

In addition, a phase III trial of Optune® (200 kHz) as monotherapy compared to active chemotherapy in recurrent glioblastoma patients showed TTFields to be equivalent to active chemotherapy in extending survival, associated with minimal toxicity, good quality of life, and activity within the brain (14% response rate). Finally, a phase III trial of Optune® combined with maintenance temozolomide compared to maintenance temozolomide alone has shown that combined therapy led to a significant improvement in both progression free survival and overall survival in patients with newly diagnosed glioblastoma without the addition of high grade toxicity and without decline in quality of life.

DESCRIPTION OF THE TRIAL:

All patients included in this trial are patients with unresectable Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma. In addition, all patients must meet all eligibility criteria.

All eligible patients will receive continuous Tumor Treating Fields (TTFields) - NovoTTF-100L (P) treatment at 150 KHz frequency, and XELOX regimen (combination of oxaliplatin + capecitabine). Patients will be assessed once every 9 weeks according to RECIST v1.1. Study treatment should be continued until disease progression, intolerable toxicity or withdrawal of informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to and be able to sign an informed consent form
2. Male or female aged ≥ 18 years
3. Be able to receive the treatment in compliance with the study protocol in the discretion of the investigator
4. ECOG Performance status score 0 or 1
5. Histologically confirmed unresectable, locally advanced or metastatic Gastroesophageal Junction (GEJ) or Gastric (GC) Adenocarcinoma. The subject must be previously untreated with systemic treatment (including chemotherapy, targeted therapy, and Onco-Immunotherapy), and without resection of primary gastric focus.
6. Subjects must have at least one measurable lesion as per RECIST 1.1 criteria; and the tumor assessment baseline should be performed and established by the investigator within 28 days prior to study treatment.
7. Life expectancy ≥ 3 months
8. The allowed previous treatment: Palliative radiotherapy for bone metastasis is allowed if it has been completed within 2 weeks prior to the study treatment and all treatment-related toxicity should be recovered to Grade 1 before enrollment, according to CTCAE 5.0.
9. Women of childbearing potential must have a negative serum pregnancy test result during screening. Post-menopausal women and surgically sterilized women are not required to undergo a pregnancy test. Females of childbearing potential/males and its partners who are sexually active must agree to adopt methods of contraception from signing the ICFs to within at least 6 months after the last dose of study drug. Besides, male subjects must be willing to refrain from sperm donation during this time.
10. Able to operate the NovoTTF-100L (P) System independently or with the help of a caregiver.

Exclusion Criteria:

1. White blood cell count (WBC) < 2 × 10^9 / L
2. Absolute neutrophil count (ANC) < 1.5 × 10^9 / L
3. Platelet count < 100 × 10^9 / L
4. Hemoglobin < 90 g/L
5. Serum albumin < 30 g/L
6. Serum creatinine > 1.5 × ULN, or creatinine clearance< 60 mL/min/1.73 m^2 calculated by Cockcroft-Gault
7. Serum total bilirubin > 1.5 × ULN
8. AST, ALT, ALP:

   1. Patients without liver metastasis or bone metastases i. AST or ALT >1.5 × ULN and ALP > 2.5 × ULN ii. AST or ALT >2.5 × ULN
   2. Patients with liver metastasis and without bone metastases i. AST or ALT > 5 × ULN and ALP > 2.5 × ULN
   3. Patients with liver metastasis and bone metastases i. AST or ALT > 5 × ULN and ALP > 10 × ULN
   4. Patients without liver metastasis and with bone metastases i. AST or ALT > 1.5 × ULN and ALP > 10 × ULN
9. Coagulation function: International Normalized Ratio (INR) > 2.3 or Prothrombin Time (PT) of > 6 seconds above the reference.
10. The other abnormal laboratory test:

    1. Electrolyte disorder including hyponatremia, hypokalemia and hypophosphatemia before the first dose, which cannot be restored by fluid and electrolyte therapies;
    2. HIV positive;
11. Metastases to central nervous system with clinical symptoms. Patients who previously received treatments for the metastases to central nervous system, are stable and meet the following requirements are allowed to be enrolled:

    1. No treatment for the metastases to central nervous system during the screening period (e. g. surgery, radiotherapy, corticosteroid therapy-prednisolone > 10 mg/day or equivalent)
    2. No progress in central nervous system lesions as indicated by MRI or CT within 14 days prior to the study treatment
    3. No meningeal metastasis or spinal cord compression
12. Moderate or severe ascites defined by physical examination and/or CT confirmed
13. Non-healing wound or ulcer within 3 months prior to study enrollment, or history of bone fracture
14. Previous allogeneic organ transplantation or allogeneic bone marrow transplantation
15. Implantable electronic medical devices in the torso.
16. Peripheral neuropathy ≥ Grade 2 (CTCAE 5.0)
17. Except hearing loss, alopecia and fatigue, all toxic reactions caused by previous anti-tumor therapy > Grade 1 (CTCAE 5.0)
18. Other malignant tumors have occurred over the past five years, with the exception of locally curable cancers treated with radical therapy, such as basal or squamous cell skin cancer, superficial bladder cancer, or in situ carcinoma of the cervix, prostate or breast.
19. Subjects who are at increased risk of bleeding or thrombosis:

    1. Clinically significant bleeding within 3 months prior to screening or clear bleeding tendency;
    2. Gastrointestinal hemorrhage within 3 months prior to screening or clear tendency of gastrointestinal hemorrhage;
    3. Arterial/venous thromboembolic events within 6 months prior to screening, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, etc.;
    4. Require anticoagulation therapy with an agent such as warfarin or heparin;
    5. Require chronic anti-platelet therapy (such as aspirin≥100 mg/day, clopidogrel, etc.);
20. History of cardiovascular disease:

    1. NYHA (New York Heart Association) grade 3 and 4 congestive heart failure;
    2. Unstable angina pectoris or newly diagnosed angina pectoris or myocardial infarction within 12 months prior to screening;
    3. Arrhythmias requiring medications other than β-blockers;
    4. Patients with valvular heart disease of ≥ CTCAE grade 2;
    5. Hypertension inadequately controlled by drugs (systolic pressure >150 mmHg or diastolic pressure >90 mmHg);
21. The investigator considers that there may be an increased risk related to the study or study treatment, or any serious or uncontrolled systemic diseases, such as infection, diabetes, hypertension, that affect the patient's ability to receive the study treatment.
22. Treatment with systemic anticancer agents (including but not limited to chemotherapy, targeted therapy, onco-immunotherapy, and biotherapy (tumor vaccines, cytokines, or cancer related growth factors)) 14 days before the study treatment, or traditional Chinese herbal medicine or Chinese patent medicine for anti-tumor therapy 7 days prior to the treatment.
23. Patients with active chronic hepatitis B or hepatitis C, or co-infection of both, patients with hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) positive during screening who have hepatitis B virus (HBV) DNA titer > 500 IU/ mL and HCV RNA detectable can be enrolled after active hepatitis B or hepatitis C infection that requires treatment have been ruled out. During the study treatment, corresponding anti-viral treatment should be given.
24. Known history of allergies or hypersensitivities to medical adhesives, hydrogel, standard drugs used in this study or their components.
25. Known history of alcohol or drug abuse.
26. Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  Investigator-assessed objective response rate (ORR) as per RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Overall survival | 2 years
Disease control rate | 2 years
Time to progression | 2 years
Duration of response | 2 years
12 month overall survival rate | 2 years
Severity and frequency of adverse events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Background] Taphoorn MJB, Dirven L, Kanner AA, Lavy-Shahaf G, Weinberg U, Taillibert S, Toms SA, Honnorat J, Chen TC, Sroubek J, David C, Idbaih A, Easaw JC, Kim CY, Bruna J, Hottinger AF, Kew Y, Roth P, Desai R, Villano JL, Kirson ED, Ram Z, Stupp R. Influence of Treatment With Tumor-Treating Fields on Health-Related Quality of Life of Patients With Newly Diagnosed Glioblastoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):495-504. doi: 10.1001/jamaoncol.2017.5082. PMID 29392280